CLINICAL TRIAL: NCT05463107
Title: Correlation Between Various Urinary Exosomal Protein Biomarkers and Pathological Manifestation in Thyroid Follicular Neoplasm: Early and Pre-operative Diagnosis of Follicular Thyroid Cancer
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202110076RINB
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Thyroid Cancer; Follicular Thyroid Cancer
Keywords: Exosome; Urine; Biological marker; Thyroglobulin; Galactin-3
MeSH Terms: conditions — Thyroid Neoplasms; Adenocarcinoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Thyroid cancer is the most common endocrine malignancy in the world. Generally, thyroid cancer could be divided into well-differentiated and poorly-differentiated. Well-differentiated thyroid cancers usually have two different patterns, including papillary thyroid cancer and follicular thyroid cancer. Thyroid sonography is convenient to obtain repeatedly for the images of nodular goiter. However, cytology and pathology are still the golden rules to make the final diagnosis. Under the basis of sono-guided fine needle aspiration cytology, diagnosis of papillary thyroid cancer is typically using fine needle aspiration cytology based on the presentation of typical cytologic features. On the other hand, thyroid follicular lesion cannot be interpretated via cytology because the evidence of capsular invasion or vascular permeation of capsule will not be available in fine needle aspiration cytology. Surgical intervention with pathological specimens is the only pathway to make the final diagnosis. Interestingly, both patterns of well-differentiated thyroid cancer shared the same follow-up tumor marker, i.e. serum thyroglobulin. Up to date, pre-operative diagnosis of follicular thyroid cancer is still one of the unresolved issues in endocrine oncology.

DETAILED DESCRIPTION:
Thyroid cancer is one of the most popular malignancy in the past several decades all over the world. For poorly-differentiated thyroid cancer, therapeutic strategy of costly target therapy together with immune therapy will be the pivotal one because of its poor prognosis. The average 5-year relative survival rate of anaplastic thyroid cancer is only 3 to 31 % on the stage from distant metastasis to localized disease.

However, it will be very different for well-differentiated thyroid cancer, and the average 5-year relative survival rate of both thyroid papillary or follicular thyroid cancer is more than 98 %. Therefore, the most important treatment strategy for endocrinologists will consider the development of biomarkers for early diagnosis and postoperative follow-up, rather than measuring serum thyroglobulin alone, which is the only biomarker in the current medical guidelines, and there is no choice. Our research team tried to find the newer biomarker together with serum thyroglobulin for post-operative longitudinal follow-up of well-differentiated thyroid cancer in the past five years. The investigators used urinary exosomal proteins as target and did find several peptides to be helpful, including our published urinary exosomal thyroglobulin (UExTg). In Taiwan, goiter and thyroid cancer are prevalent diseases. Although papillary thyroid cancer could be diagnosed via reliable sono-guided fine needle aspiration cytology, follicular thyroid cancer is still an unresolved issue in daily medical practice, especially in cytology. the investigators need to find a practicably earlier biomarker, which should be convenient, non-invasive and repeatable in sample collection. In our previous research and published data, urine will be a reliable source of data.

Exosomes are nano-vesicles, containing DNA, RNA and proteins, and usually secreted by cells into extracellular spaces. Generally, the vesicles of exosomes are only 40 to 150 nm in diameter. Exosomes may carry and transfer the messages between different tissues. Now, the existing evidences revealed that exosomes may represent certain messages from malignant cells, including diagnosed biomarkers or prognostic predictors. Previously, published data of exosomal studies in thyroid cancer focused on serum microRNA, long coding RNA and circular RNA, but only few published data on peptides, which were named as liquid biopsy. However, cell-secreted exosomes of malignancy could be collected not only in plasma, body fluid, but also from urine, which is the non-invasive pathway but valuable wastes of human body. Our research group had developed experienced technique to collect urinary exosomes via our pilot study in the past several years.

Since the investigators proved the role of urinary exosomal thyroglobulin, UExTg, in post-operative follow-up in well-differentiated thyroid cancer in the past three years, from 2018-2020, the investigators also found several peptides to be the candidates of prognostic predictors in our preliminary studies, including Calprotectin A8/A9, Annexin-2, Angiopoietin-1.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed patients with nodular goiter or multinodular goiter, thyroid papillary, follicular and anaplastic thyroid cancer, pre-operation.

Exclusion Criteria:

* unclearly diagnosed patients with thyroid papillary, follicular and anaplastic thyroid cancer

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Clinical study was designed as prospective pattern, and enrolled patients with nodular goiter or multinodular goiter, who had received fine needle aspiration cytology and/or thyroidectomy. Cytology and complete surgical pathology survey will be recorded for cytological and surgical samples. This study will enroll 50 consecutive patients with nodular goiter or multinodular goiter in 2nd and 3rd years.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Change of serum thyroglobulin level | Within 36 months
  Thyroid function test
Change of serum free T4 level | Within 36 months
  Thyroid function test
Change of serum TSH level | Within 36 months
  Thyroid function test
Change of anti-thyroglobulin level | Within 36 months
  Thyroid function test
Urinary exosomal thyroglobulin detection | Within 36 months
  Urinary exosomal biomarker
Urinary exosomal galectin-3 detection | Within 36 months
  Urinary exosomal biomarker
Urinary exosomal calprotectin A9 detection | Within 36 months
  Urinary exosomal biomarker
Urinary exosomal transketolase detection | Within 36 months
  Urinary exosomal biomarker
Urinary exosomal keratin 19 detection | Within 36 months
  Urinary exosomal biomarker
Urinary exosomal angiopoietin-1 detection | Within 36 months
  Urinary exosomal biomarker
Urinary exosomal tissue inhibitor of metalloproteinase detection | Within 36 months
  Urinary exosomal biomarker
Urinary exosomal keratin 8 detection | Within 36 months
  Urinary exosomal biomarker
Urinary exosomal calprotectin A8 detection | Within 36 months
  Urinary exosomal biomarker
Urinary exosomal annexin II detection | Within 36 months
  Urinary exosomal biomarker
Urinary exosomal afamin detection | Within 36 months
  Urinary exosomal biomarker

SECONDARY OUTCOMES:
Thyroid fine needle aspiration cytology | Within 36 months
  Urinary exosomal biomarker
Ultrasonography of thyroid nodules | Within 36 months
  Urinary exosomal biomarker

CONTACTS AND LOCATIONS:
Overall Officials: CHIH-YUAN WANG, Doctor, Principal Investigator — Department of Internal Medicine, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan